CLINICAL TRIAL: NCT02703038
Title: French Observatory on the Management of Cardiogenic Shock in 2016
Acronym: FRENSHOCK
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 15897
Record Dates: First submitted 2016-02-23; First posted 2016-03-09 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Shock, Cardiogenic
Keywords: cardiogenic shock; observatory
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiogenic shock: Patient with cardiogenic shock table defined by the combination of a low cardiac output even as the filling pressures are normal or high, originally of hypoperfusion and organ suffering.

SUMMARY:
Cardiogenic shock (CS) is defined as an organ hypoperfusion secondary to low cardiac output. Catches diagnostic management, and therapeutic monitoring of these patients remain highly variable from one center to another and even from one doctor to another within the same team. The management protocols are often not standardized or non-existent.

It appears therefore necessary to make an inventory of the management practices of the CS in France in 2016, prerequisite to a common work of standardization of practices and the creation of specialized networks to support these complex patients.

DETAILED DESCRIPTION:
The Observatory FRENSHOCK proposes to set up a cohort of 500 patients recruited prospectively over a period of 6 months.

Patients will be followed up at 1 month and 1 year Patients should have agreed to participate in the observatory, knowing that participation or refusal to participate will not alter the therapeutic attitude of the physician responsible for the patient. The study of phenotypic characteristics will not change the therapeutic approach of the medical teams.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Cardiogenic shock authenticated by the existence of at least one positive test for each of the following three parts:

(A) Low cardiac output (1 criterion necessary and sufficient):

* Clinic: SBP <90mmHg and / or need to maintain inotropic or vasopressor to maintain SBP> 90 mmHg
* Echocardiography: IC <2.2L / min / m2 and / or LVEF <30%
* Hemodynamics by Swan Ganz catheterization or right: IC 2.2 l / min / m2 (B) elevation of pulmonary pressure / left surcharge (1 criterion necessary and sufficient):
* Clinical (IVD and abortion);
* Radiological (Surcharge on RT or chest CT);
* Organic (NTproBNP> 900pg / ml or BNP> 400pg / ml);
* Echocardiography (E / A> 2 if LVEF <45% or E / Ea> 13 if normal LVEF, or PAPS> 35mmHg and / or TDE <150ms and / or Ap-Am> 30ms and / or E / 2 Vp≥ , 5);
* Right Swan Ganz catheterization or (pulmonary capillary pressures> 15mmHg and / or mPAP> 25mmHg)

(C) Organs malperfusion (1 criterion necessary and sufficient):

* Clinic: oliguria <30ml / kg / h, mottling, consciousness disorders)
* Organic: arterial lactate> 2 mmol / L, liver failure, kidney failure

Exclusion Criteria:

* Final diagnosis retained other than cardiogenic shock
* Cardiac arrest without spontaneous activity in the hospital management
* Post-cardiotomy cardiogenic shock
* Deprived of liberty patient
* Refusal or lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (> 18 years) with cardiogenic shock table defined by the combination of a low cardiac output even as the filling pressures are normal or high, originally of hypoperfusion and suffering of organ.
Sampling Method: Non-Probability Sample
Enrollment: 777 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Mortality at day 30 | 30 days
  Death rate at 30 days of follow-up

SECONDARY OUTCOMES:
Analysis of mortality at day 30 by subgroup on age, sex, NYHA grade, initial etiology | 30 days
  Rate of mortality at day 30 distributed by subgroup on age, sex, NYHA grade, initial etiology (Including ischemic versus non-ischemic heart disease, type and assistance and medical treatment)
Mortality at 1 year | 1 year
  Death rate at 1 year of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Clément DELMAS, Principal Investigator — AP
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reynolds HR, Hochman JS. Cardiogenic shock: current concepts and improving outcomes. Circulation. 2008 Feb 5;117(5):686-97. doi: 10.1161/CIRCULATIONAHA.106.613596. No abstract available. PMID 18250279
- [Background] Aissaoui N, Puymirat E, Tabone X, Charbonnier B, Schiele F, Lefevre T, Durand E, Blanchard D, Simon T, Cambou JP, Danchin N. Improved outcome of cardiogenic shock at the acute stage of myocardial infarction: a report from the USIK 1995, USIC 2000, and FAST-MI French nationwide registries. Eur Heart J. 2012 Oct;33(20):2535-43. doi: 10.1093/eurheartj/ehs264. Epub 2012 Aug 26. PMID 22927559
- [Background] Jeger RV, Radovanovic D, Hunziker PR, Pfisterer ME, Stauffer JC, Erne P, Urban P; AMIS Plus Registry Investigators. Ten-year trends in the incidence and treatment of cardiogenic shock. Ann Intern Med. 2008 Nov 4;149(9):618-26. doi: 10.7326/0003-4819-149-9-200811040-00005. PMID 18981487
- [Background] Thiele H, Allam B, Chatellier G, Schuler G, Lafont A. Shock in acute myocardial infarction: the Cape Horn for trials? Eur Heart J. 2010 Aug;31(15):1828-35. doi: 10.1093/eurheartj/ehq220. Epub 2010 Jul 7. PMID 20610640
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, de Waha A, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Lauer B, Bohm M, Ebelt H, Schneider S, Werdan K, Schuler G; Intraaortic Balloon Pump in cardiogenic shock II (IABP-SHOCK II) trial investigators. Intra-aortic balloon counterpulsation in acute myocardial infarction complicated by cardiogenic shock (IABP-SHOCK II): final 12 month results of a randomised, open-label trial. Lancet. 2013 Nov 16;382(9905):1638-45. doi: 10.1016/S0140-6736(13)61783-3. Epub 2013 Sep 3. PMID 24011548
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Fuhrmann J, Bohm M, Ebelt H, Schneider S, Schuler G, Werdan K; IABP-SHOCK II Trial Investigators. Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1287-96. doi: 10.1056/NEJMoa1208410. Epub 2012 Aug 26. PMID 22920912
- [Background] Sleeper LA, Reynolds HR, White HD, Webb JG, Dzavik V, Hochman JS. A severity scoring system for risk assessment of patients with cardiogenic shock: a report from the SHOCK Trial and Registry. Am Heart J. 2010 Sep;160(3):443-50. doi: 10.1016/j.ahj.2010.06.024. PMID 20826251
- [Background] Katz JN, Stebbins AL, Alexander JH, Reynolds HR, Pieper KS, Ruzyllo W, Werdan K, Geppert A, Dzavik V, Van de Werf F, Hochman JS; TRIUMPH Investigators. Predictors of 30-day mortality in patients with refractory cardiogenic shock following acute myocardial infarction despite a patent infarct artery. Am Heart J. 2009 Oct;158(4):680-7. doi: 10.1016/j.ahj.2009.08.005. PMID 19781431
- [Background] Thiele H, Ohman EM, Desch S, Eitel I, de Waha S. Management of cardiogenic shock. Eur Heart J. 2015 May 21;36(20):1223-30. doi: 10.1093/eurheartj/ehv051. Epub 2015 Mar 1. PMID 25732762
- [Background] De Backer D, Biston P, Devriendt J, Madl C, Chochrad D, Aldecoa C, Brasseur A, Defrance P, Gottignies P, Vincent JL; SOAP II Investigators. Comparison of dopamine and norepinephrine in the treatment of shock. N Engl J Med. 2010 Mar 4;362(9):779-89. doi: 10.1056/NEJMoa0907118. PMID 20200382
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Mebazaa A, Nieminen MS, Packer M, Cohen-Solal A, Kleber FX, Pocock SJ, Thakkar R, Padley RJ, Poder P, Kivikko M; SURVIVE Investigators. Levosimendan vs dobutamine for patients with acute decompensated heart failure: the SURVIVE Randomized Trial. JAMA. 2007 May 2;297(17):1883-91. doi: 10.1001/jama.297.17.1883. PMID 17473298
- [Background] Felker GM, Benza RL, Chandler AB, Leimberger JD, Cuffe MS, Califf RM, Gheorghiade M, O'Connor CM; OPTIME-CHF Investigators. Heart failure etiology and response to milrinone in decompensated heart failure: results from the OPTIME-CHF study. J Am Coll Cardiol. 2003 Mar 19;41(6):997-1003. doi: 10.1016/s0735-1097(02)02968-6. PMID 12651048
- [Background] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Background] Dzavik V, Sleeper LA, Cocke TP, Moscucci M, Saucedo J, Hosat S, Jiang X, Slater J, LeJemtel T, Hochman JS; SHOCK Investigators. Early revascularization is associated with improved survival in elderly patients with acute myocardial infarction complicated by cardiogenic shock: a report from the SHOCK Trial Registry. Eur Heart J. 2003 May;24(9):828-37. doi: 10.1016/s0195-668x(02)00844-8. PMID 12727150
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] O'Connor CM, Gattis WA, Uretsky BF, Adams KF Jr, McNulty SE, Grossman SH, McKenna WJ, Zannad F, Swedberg K, Gheorghiade M, Califf RM. Continuous intravenous dobutamine is associated with an increased risk of death in patients with advanced heart failure: insights from the Flolan International Randomized Survival Trial (FIRST). Am Heart J. 1999 Jul;138(1 Pt 1):78-86. doi: 10.1016/s0002-8703(99)70250-4. PMID 10385768
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL. 2013 ACCF/AHA guideline for the management of heart failure: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):1810-52. doi: 10.1161/CIR.0b013e31829e8807. Epub 2013 Jun 5. No abstract available. PMID 23741057
- [Result] Delmas C, Puymirat E, Leurent G, Elbaz M, Manzo-Silberman S, Bonello L, Gerbaud E, Bataille V, Levy B, Lamblin N, Bonnefoy E, Henry P, Roubille F; FRENSHOCK investigators. Design and preliminary results of FRENSHOCK 2016: A prospective nationwide multicentre registry on cardiogenic shock. Arch Cardiovasc Dis. 2019 May;112(5):343-353. doi: 10.1016/j.acvd.2019.02.001. Epub 2019 Apr 11. PMID 30982720
- [Derived] Cherbi M, Roubille F, Gerbaud E, Bonnefoy E, Lamblin N, Bonello L, Levy B, Lim P, Merdji H, Elbaz M, Khachab H, Bourenne J, Seronde MF, Schurtz G, Harbaoui B, Vanzetto G, Combaret N, Lattuca B, Leurent G, Puymirat E, Delmas C. Clinical profile, short and long-term outcomes of non-ischaemic cardiogenic shock: A FRENSHOCK sub-analysis. ESC Heart Fail. 2025 Jun;12(3):2335-2346. doi: 10.1002/ehf2.15046. Epub 2025 Mar 25. PMID 40130820
- [Derived] Volle K, Merdji H, Bataille V, Lamblin N, Roubille F, Levy B, Champion S, Lim P, Schneider F, Labbe V, Khachab H, Bourenne J, Seronde MF, Schurtz G, Harbaoui B, Vanzetto G, Quentin C, Combaret N, Marchandot B, Lattuca B, Biendel C, Leurent G, Bonello L, Gerbaud E, Puymirat E, Bonnefoy E, Aissaoui N, Delmas C; FRENSHOCK Investigator. Ventilation strategies in cardiogenic shock: insights from the FRENSHOCK observational registry. Clin Res Cardiol. 2025 Oct;114(10):1311-1323. doi: 10.1007/s00392-024-02551-x. Epub 2024 Oct 23. PMID 39441346
- [Derived] Roubille F, Cherbi M, Kalmanovich E, Delbaere Q, Bonnefoy-Cudraz E, Puymirat E, Schurtz G, Gerbaud E, Bonello L, Lim P, Leurent G, Roubille C, Delmas C. The admission level of CRP during cardiogenic shock is a strong independent risk marker of mortality. Sci Rep. 2024 Jul 16;14(1):16338. doi: 10.1038/s41598-024-67556-y. PMID 39014136
- [Derived] Manzo-Silberman S, Martin AC, Boissier F, Hauw-Berlemont C, Aissaoui N, Lamblin N, Roubille F, Bonnefoy E, Bonello L, Elbaz M, Schurtz G, Morel O, Leurent G, Levy B, Jouve B, Harbaoui B, Vanzetto G, Combaret N, Lattucca B, Champion S, Lim P, Bruel C, Schneider F, Seronde MF, Bataille V, Gerbaud E, Puymirat E, Delmas C; FRENSHOCK investigators. Sex disparities in cardiogenic shock: Insights from the FRENSHOCK registry. J Crit Care. 2024 Aug;82:154785. doi: 10.1016/j.jcrc.2024.154785. Epub 2024 Mar 16. PMID 38493531
- [Derived] Cherbi M, Bouisset F, Bonnefoy E, Lamblin N, Gerbaud E, Bonello L, Levy B, Lim P, Joffre J, Beuzelin M, Roland Y, Niquet L, Favory R, Khachab H, Harbaoui B, Vanzetto G, Combaret N, Marchandot B, Lattuca B, Leurent G, Lairez O, Puymirat E, Roubille F, Delmas C. Characteristics, management, and mid-term prognosis of older adults with cardiogenic shock admitted to intensive care units: Insights from the FRENSHOCK registry. Int J Cardiol. 2024 Jan 15;395:131578. doi: 10.1016/j.ijcard.2023.131578. Epub 2023 Nov 11. PMID 37956759
- [Derived] Cherbi M, Bonnefoy E, Lamblin N, Gerbaud E, Bonello L, Roubille F, Levy B, Champion S, Lim P, Schneider F, Elbaz M, Khachab H, Bourenne J, Seronde MF, Schurtz G, Harbaoui B, Vanzetto G, Combaret N, Labbe V, Marchandot B, Lattuca B, Biendel-Picquet C, Leurent G, Puymirat E, Maury P, Delmas C. One-year outcomes in cardiogenic shock triggered by supraventricular tachycardia: an analysis of the FRENSHOCK multicenter prospective registry. Front Cardiovasc Med. 2023 Sep 5;10:1167738. doi: 10.3389/fcvm.2023.1167738. eCollection 2023. PMID 37731529
- [Derived] Cherbi M, Roubille F, Lamblin N, Bonello L, Leurent G, Levy B, Elbaz M, Champion S, Lim P, Schneider F, Cariou A, Khachab H, Bourenne J, Seronde MF, Schurtz G, Harbaoui B, Vanzetto G, Quentin C, Delabranche X, Aissaoui N, Combaret N, Tomasevic D, Marchandot B, Lattuca B, Henry P, Gerbaud E, Bonnefoy E, Puymirat E, Maury P, Delmas C. One-year outcomes in cardiogenic shock triggered by ventricular arrhythmia: An analysis of the FRENSHOCK multicenter prospective registry. Front Cardiovasc Med. 2023 Jan 26;10:1092904. doi: 10.3389/fcvm.2023.1092904. eCollection 2023. PMID 36776263